# Penn Medicine Research Participant

## Combined Informed Consent Form and HIPAA Authorization

Protocol Title: PARPVAX2: A Phase II Study of Maintenance Niraparib Plus Ipilimumab

in Patients with Metastatic Pancreatic Cancer Whose Disease Has Not

Progressed on Platinum-Based Chemotherapy

**Collaborators:** The Lustgarten Foundation, Bristol-Myers Squibb (BMS),

GlaxoSmithKline (GSK), and Dana Farber Cancer Institute

Regulatory Sponsor: University of Pennsylvania

Principal Investigator: Kim A. Reiss, MD

Abramson Cancer Center of the University of Pennsylvania

Philadelphia, PA 19104

215-360-0735

**Sub-investigators:** Mark O'Hara, MD; Ursina Teitelbaum, MD; Charles Schneider, MD; Ryan

Massa, MD; Jennifer Eads, MD, Parul Agarwal, MD; William Chapin, MD

**Emergency Contact:** 24 Hour Emergency – Call 215-662-4000

Ask for Oncologist On-Call

# **Summary**

You are being invited to participate in a research study. Your participation is voluntary, and you should only participate if you completely understand what the study requires and what the risks of participation are. You should ask the study team any questions you have before agreeing to join the study. If you have any questions about your rights as a human research participant at any time before, during or after participation, please contact the Institutional Review Board (IRB) at (215) 898-2614 for assistance.

You are being invited to participate in a research study because you have pancreatic cancer. This research study is designed to learn more about the effectiveness of niraparib with ipilimumab given to individuals who have been diagnosed with pancreatic cancer. Your cancer may or may not improve from participating in this study. The hope is that this study treatment may provide a new treatment option for patients with pancreatic cancer, however, such a benefit cannot be guaranteed.

If you agree to join the study, you will be randomized to receive the study drugs or standard chemotherapy and be asked to complete the following research procedures: research blood tests, including a pregnancy test if you are able to bear children, and tumor biopsy. Additional procedures that are consistent with your standard of care treatment will also be performed.

Version: 1/21/2025 1 of 27

Your participation will last up to until your disease progresses or you experience side effects that require treatment be stopped. Even after you discontinue study treatment, you will be contacted in 30 days or 90 days, and then annually by a study team representative who will ask questions about your health.

The following are some of the most commonly observed side effects: with Niraparib, decreased blood cells such as white blood cells, red blood cells, and platelets, and with Ipilimumab, increased liver enzymes. There is always the possibility that unknown risks and side effects may occur. These may be mild or serious, and in some cases, may be very serious, long-lasting, or may never go away. There may also be a risk of death.

Other treatment options may be available to you. These could include treatment of your symptoms, without any effect on your disease, treatment with currently approved drugs, and/or participation in other clinical trials for pancreatic cancer. Your study doctor or regular doctor can discuss alternate treatments available for your condition, and any known risks related to these treatments.

The study drugs have been given to patients with pancreatic cancer in a previously published clinical trial and have provided some benefit, although the possible benefit to you is not guaranteed. In the prior study, patients who received niraparib and ipilimumab experienced the typical side effects of these two agents. There was no evidence that combining the agents resulted in an increased risk of toxicities from either drug You may also decide to forego further treatment. Please note that there are other factors to consider before agreeing to participate such as additional procedures, use of your personal information, costs, and other possible risks not discussed here. You are free to decline or stop participation at any time during or after the initial consenting process.

# Why am I being asked to volunteer?

You are being asked to participate in this research study because you have been diagnosed with advanced pancreatic cancer. Your participation is voluntary, which means you can choose whether or not you want to participate. If you choose not to participate, your clinical care will not be affected. Before agreeing to participate in this research study, it is important that you read the following explanation of the proposed procedures and how long you will be in the study. This document describes the purpose, procedures, benefits, risks, discomforts and precautions of the study. It also describes the alternative procedures that are available to you and your right to withdraw from the study at any time.

Please take time to read the following information carefully. You may wish to discuss it with your family, friends, and your personal doctor (i.e., your family doctor or primary care doctor). If you have any questions, you may ask your study doctor and/or the research team for more information. Take time to decide whether or not you wish to take part. If you decide to participate, you will be asked to sign this form. If you decide to participate, you can change your mind at any time and withdraw from the study without giving a reason.

# What is the purpose of this research study? What does this study involve?

The main purpose of this study is to see how well the drugs niraparib and ipilimumab work together to stop the growth of your pancreatic cancer.

Version: 1/21/2025 2 of 27

The United States Food and Drug Administration (US FDA) is an authority that regulates new medicines. The study drugs niraparib and ipilimumab are approved by the US FDA to treat certain types of cancer. However, the use of niraparib and ipilimumab in this study is investigational because these drugs are not approved to treat advanced pancreatic adenocarcinoma. However, as described above, a prior clinical trial demonstrated that niraparib and ipilimumab was effective in patients with advanced pancreatic cancer whose cancer had not grown during treatment with chemotherapy. This current study is designed to further validate that finding.

This study will involve two different treatment arms. In Arm A, patients will receive niraparib plus ipilimumab. In Arm B, patients will receive standard of care chemotherapy. Patients will be randomized to one of the two arms in a 3:1 fashion. This means that for every three patients who receive niraparib plus ipilimumab, one will receive standard chemotherapy

## Who is sponsoring this study?

Dr. Kim A. Reiss, the Principal Investigator, is also the sponsor (entity responsible for the design, conduct and regulatory oversight of the study). GSK is the manufacturer of the study drug, niraparib, and will be providing the drug during this research study. BMS is the manufacturer of the study drug, ipilimumab, and will be providing the drug during this research study. Dr. Kim A. Reiss and Penn Medicine will receive payments to cover some of the research costs such as the collecting/reporting study information associated with the conduct of the study.

# How long will I be in the study?

You may remain on the study treatment for as long as you are benefiting from it. You may continue to participate on this study until your disease gets worse, you experience unacceptable side effects, and/or your physician no longer believes the therapy is of benefit to you (whichever occurs first).

Once you stop the study drug treatments, there will be an End of Treatment visit and a 30-day follow-up visit. After your 30-day follow-up visit you will be followed for safety up to 90 days. Then the study team will contact you annually by telephone, email, monitor your medical records, or at your clinical visits to ask you questions about your health. You may stop your participation in the study at any time.

# What am I being asked to do?

If you meet all of the criteria for being in the study, you will be registered to participate. The study procedures are outlined below.

<u>Screening Procedures:</u> These procedures are done to evaluate your cancer, overall health, and eligibility. If you have had some of these tests/procedures recently, they may not need to be repeated. These tests and procedures need to be done within 28 days before you receive your first dose of study drugs, unless otherwise indicated.

The following procedures are being performed as part of your participation in the research study:

Version: 1/21/2025 3 of 27

- Blood sample (about 1 teaspoon of blood) for HIV viral status testing to check if you have these viruses. This is to ensure you are healthy enough to enter the study.
- Research biopsies of your cancer at two time points during your participation on the trial
- Blood samples (about 5 tablespoons of blood) taken for research analyses at various time points during your participation on the trial
- You must agree not to donate blood during your participation and for 90 days after the last dose of treatment.

The following procedures are part of your standard care and would be performed regardless of your participation in the research study:

- A complete physical examination including height and weight.
- A review of your history to include: a review of your medical and cancer history to make sure you do not have any conditions that could interfere with your taking part in this study (this will include the review of results from genetic testing you have already had); you will be asked how you are feeling; a review of the medications you are taking, including all prescription medications and all non-prescription medications (such as vitamins, herbal supplements, aspirin, etc.); a review of your social history (such as if you are a smoker and how much alcohol you may drink); and a review of any significant medical or surgical procedures you have had.
- Your demographic information will be captured which include your gender, age, race, and ethnicity.
- An assessment of how your disease affects your daily living abilities (called Performance Status).
- Measurement of your vital signs (blood pressure, pulse, and temperature).
- Approximately 2 tablespoons of blood will be drawn to determine your eligibility. The routine tests being done to determine your eligibility and for safety purposes will test your blood cell counts (number of each type of blood cell), blood chemistry levels (to test your kidney and liver function and the minerals in your body), test for thyroid gland problems and a serum pregnancy test for women of childbearing potential. If the pregnancy test comes back positive you will not be allowed to participate in this study.
- Radiology tests to assess your disease. These assessments may include a CT (computed tomography) scan, MRI (magnetic resonance imaging) scan, PET/CT (positron emission tomography/computed tomography) scan, and/or a chest x-ray.

Once you have passed the screening, but before you begin receiving study drug, the following may be performed:

- If you have stored tumor tissue available from a previous biopsy, this will be documented and
  we will collect some of the stored tumor tissue for research testing prior to conclusion of the
  study.
  - This would not typically be done as a part of your standard of care treatment.
- If you have a tumor that can easily be reached, you will be asked to allow your doctor to complete two tumor biopsies and remove a small amount of tumor. This is a required part of this study (is not optional) if the biopsy is feasible. Providing this type of tumor sample is

Version: 1/21/2025 4 of 27

essential in helping us learn about your specific disease and how we can help other patients like you.

o This would not typically be done as a part of your standard of care treatment.

## Procedures associated with the administration of the study drug(s)

When all of the above tests/procedures have been completed, if you have been found to be eligible to enter this study, and you agree to participate, you will be randomized to treatment Arm A or Arm B and be scheduled to receive the study drugs.

Study drugs will be given over many cycles. A cycle is the time between the start of 1 round of treatment until the start of the next round. In this study, Arm A with Niraparib plus Ipilimumab treatment cycle is 21 days and Arm B with standard of care medication is 28 days. Cycles will continue until your cancer gets worse, you experience unacceptable side effects, your doctor no longer believes the therapy is in your best interest, or you no longer want to participate in the study.

In this study, a process called randomization will be used to determine who will receive Niraparib plus ipilimumab OR standard of care chemotherapy (FOLFIRI). Randomization is when participants are randomly put into different groups in a study. Three of four patients will receive Niraparib plus ipilimumab.

Your doctor and the study team will inform you if you will receive Niraparib plus ipilimumab OR a standard of care medication. Ipilimumab will be administered during your scheduled visit and all patients will be given a diary to document that the study medication, niraparib, will be taken at home between visits. You will be asked to bring this completed diary and your remaining study drug and/or empty pill bottles to each study visit. When you return the study drug bottles and diary, the study team will review everything to make sure you are taking the drug appropriately and completing this diary as requested.

If you are randomized to receive niraparib plus ipilimumab (Arm A), treatment is as follows beginning on Day 1 of each 21 day cycle:

- Niraparib two 100 mg pills by mouth (oral) daily
- Ipilimumab 30 minute (IV, into a vein) infusion on day 1 of the first 4 cycles. Niraparib will continue after you have stopped ipilimumab.

If you are randomized to receive a standard of care medication (Arm B), treatment is as follows beginning on Day 1 of each 28 day cycle:

FOLFIRI 30 minutes (IV, into a vein) infusion on day 1 and 15 of every cycle.

#### Study Tests/Procedures following Screening

These exams, tests, and procedures are being done to evaluate your health and response to the study drug(s). At each of these study visits you will be asked how you are feeling, if you have had any side effects, if you may be pregnant, if you have had any medical procedures, and about any medications you are taking. It is important you check with your study doctor before starting any new medications. Taking other drugs (including alcohol, over-the-counter medications, herbal preparations, illegal drugs, or Version: 1/21/2025

nutritional supplements) may cause additional side effects or even life-threatening reactions when combined with the drugs being used in this study. If you experience side effects, changes in your health and/or changes in medications, please contact your study doctor or a study team member.

You will have the following tests, procedures, and assessments done at the time points below:

| Arm A Schedule | | |
|---|---|---|
| Procedure/ Study Day | Day 1 of each cycle <sup>7</sup> | Weekly |
| Physical Exam, Weight | X | |
| Performance Status Evaluation | X | |
| Vital Signs | X | |
| Blood Pressure Monitoring | X | X <sup>5</sup> |
| Safety Blood Tests – about 2 tablespoons will | X | Х |
| be collected <sup>4</sup> | | |
| Research Blood Tests – about 5 tablespoons | X <sup>6</sup> | |
| will be collected <sup>1</sup> | | |
| Pregnancy Blood Test | X | |
| Review of Adverse Events | X | |
| Review of Concomitant Medications and | X | |
| Procedures | | |
| Disease Assessment/Tumor Scans <sup>2</sup> | X | |
| Tumor Biopsy <sup>3</sup> | X | |

- 1. This procedure would not typically be done as a part of standard of care treatment. We will collect research blood tests every other cycle or every 8 weeks.
- 2. Tumor scans to be performed within 7 days prior to start of every 3rd cycle or approximately every 9 weeks.
- 3. A tumor biopsy will be performed at Cycle 4 day 1 unless it is deemed unsafe by the study doctor or if there appears to be no evidence of disease (complete remission)
- 4. For safety purposes you will have a blood test for blood cell counts (number of each type of blood cell) once a week during the first 4 weeks on treatment
- 5. You will be required to take your blood pressure once every week during the first 2 months you are taking Niraparib and record this information on your study drug diary. This will also be taken at the start of each cycle while you are participating.
- 6. An additional research blood draw may be performed on day 8 of Cycle 1.
- 7. Patients on Arm A who are stable (as per the investigator) following 17 full cycles of treatment may go twelve weeks (i.e. four cycles) between clinical assessments and disease assessment imaging. For these patients, four cycles of niraparib may be dispensed at one time. However, all safety blood work must still be collected at D1 (+/- 3 days) of each cycle and will be reviewed by the research team.

| Arm B Schedule | |
|-----------------------------------------------|---------------------|
| Procedure/ Study Day | Day 1 of each cycle |
| Physical Exam, Weight | Х |
| Performance Status Evaluation | X |
| Vital Signs | X |
| Safety Blood Tests – about 2 tablespoons will | Х |
| be collected <sup>4</sup> | |

Version: 1/21/2025 6 of 27

| Research Blood Tests – about 5 tablespoons | X <sup>5</sup> |
|---------------------------------------------|----------------|
| will be collected <sup>1</sup> | |
| Review of Adverse Events | X |
| Review of Concomitant Medications and | X |
| Procedures | |
| Disease Assessment/Tumor Scans <sup>2</sup> | X |
| Tumor Biopsy <sup>3</sup> | X |

- 1. This procedure would not typically be done as a part of standard of care treatment. We will collect research blood tests every other cycle or every 8 weeks.
- 2. Tumor scans to be performed within 7 days prior to start of every 3rd cycle or approximately every 9 weeks.
- 3. A tumor biopsy will be performed at Cycle 4 day 1 unless it is deemed unsafe by the study doctor or if there appears to be no evidence of disease (complete remission)
- 4. For safety purposes you will have a blood test for blood cell counts (number of each type of blood cell) once a week during the first 4 weeks on treatment
- 5. An additional research blood draw may be performed on day 8 of Cycle 1.

## End of Study Visit:

The following procedures will be performed for all patients as soon as possible after the last dose of study treatment:

- A complete physical examination including weight
- You will be asked how you are feeling, if you have had any side effects, if you may be pregnant, if you have had any medical procedures, and about any medications you are taking.
- An assessment of how your disease affects your daily living abilities (called Performance Status)
- Measurement of your vital signs (blood pressure, pulse, and temperature)
- Approximately 6 tablespoons of blood will be drawn
  - The routine tests being done will test your blood cell counts (number of each type of blood cell), blood chemistry levels (to test your kidney and liver function and the minerals in your blood), and markers of cancer in your blood (CA19-9 and/or CEA).
  - The research tests being done to detect potential markers of clinical response to treatment, such as various types of white blood cells and their activation status. This would not typically be done as a part of your standard of care treatment.
- Radiology tests to assess your disease. These assessments may include a CT scan, MRI scan and/or PET/CT scan.
- If you are randomized to receive niraparib plus ipilimumab (Arm A), you will have a review of all
  niraparib tablets you brought back to the study center and a review of your completed study
  drug dosing diary.

#### Post-Study Procedures:

You will be asked to come in again 30 days after you have finished study treatment for a review of your general health and to see whether anything new has happened to you since your last study visit, including

Version: 1/21/2025 7 of 27

any side effects you may be experiencing.

- Report any changes in health (including any side effects)
- Radiology tests to assess your disease. These assessments may include a CT scan, MRI scan, PET/CT scan, and/or a chest x-ray (if not already done for End of Treatment visit)

After this visit, If you are randomized on Arm A, the study staff will continue to follow up with you for up to 90 days for safety. Then the study team will contact you annually by telephone, email, medical record review, or at a clinic visit to see how you are doing.

## What are the possible risks or discomforts?

While on the study, you are at risk for the following side effects. Some of these side effects may be potentially serious or life-threatening, and may include death. You should discuss these with the study doctor. There also may be other side effects that are not known and other very rare side effects that are known but not included in this list. If you experience side effects from the study drug(s), your study doctor may delay or skip a dose of the study drug, or ask you to stop taking study drug. Your doctors may also give you other drugs to help lessen these side effects. Many side effects go away shortly after the study drug is stopped, but in some cases side effects can be serious, long lasting or permanent.

Clinical studies have shown that using niraparib in combination with ipilimumab in pancreatic cancer does not increase side effects of either drug as compared to using these drugs alone.

#### **Niraparib**

The treatment with niraparib could result in side effects. The frequencies below are based on niraparib clinical trials.

Niraparib has moderate influence on the ability to drive or use machines. Patients who take niraparib may experience weakness, fatigue, difficulty concentrating and dizziness. Patients who experience these symptoms should observe caution when driving or using machines.

Known side effects of niraparib are listed below:

#### Very Common occurrence (may affect more than 1 in 10 people)

- Decrease in blood cells (red blood cells) that carry oxygen; this may make you feel tired or short of breath
- Decrease in blood cells (platelets) that help stop bleeding; this may increase your risk of bleeding
- Decrease in neutrophils, one of several types of white blood cells that fight infection; this may decrease your ability to fight infections
- Decrease in the number of white blood cells that fight infection
- Increased blood pressure
- Noticeably rapid, strong, or irregular heartbeat
- Infrequent hard stools (constipation)

Version: 1/21/2025 8 of 27

- Feeling sick to your stomach
- Vomiting
- Feeling not hungry; decreased appetite
- Sleeplessness, trouble sleeping
- Headache
- Feeling tired, lack of energy
- Shortness of breath
- Runny or stuffy nose
- Cough
- Feeling abnormal physical weakness or lack of energy
- Dizziness
- Joint pain
- Back pain
- Stomach pain
- Indigestion
- Frequent watery stools (diarrhea)
- Painful and frequent urination

#### Common occurrence (may affect up to 1 in 10 people):

- An abnormally rapid heart rate
- Infection due to low white blood cell counts
- Low blood cell counts due to a problem in the bone marrow or blood cancer starting from the bone marrow
- An irritation or infection in the tubes that carry air in and out of the lungs, that causes a cough
- Swelling of lower legs and feet
- Muscle pain
- Rash
- Decrease in weight
- Feelings of sadness, depressed (depression)
- Feelings of worry, nervousness or unease (anxiety)
- Impaired concentration, understanding, memory, and thinking
- Inflammation of the eye
- Nose bleed
- Sore, red mouth
- Swelling or irritation of the lining of the mouth, throat, esophagus, stomach or intestines
- Abnormal taste in mouth
- Dry mouth
- Increased sensitivity of the skin to sunlight
- Decrease in potassium in the blood
- Increased level of creatinine in your blood, which may be a sign of kidney damage

Version: 1/21/2025 9 of 27

- Increased levels of substances in the blood produced by the liver, which may be a sign of liver injury
- Other abnormal labs (alkaline phosphatase [ALP] increased)
- Allergic reaction, including anaphylaxis

## <u>Uncommon Occurrence (may affect up to 1 in 100 people):</u>

- Fever with low white blood cell count
- Severe life-threatening infection due to low white cell counts (associated with low blood pressure and possible organ failure (for example, heart, kidney and/or liver)
- Decrease in number of all types of blood cells
- Confusion
- Seeing or hearing things that are not likely there (hallucination)
- Inflammation of the lungs which can cause shortness of breath and difficulty breathing

## Rare Occurrence (may affect up to 1 in 1000 people):

- Severe increase in blood pressure
- A brain condition with symptoms including seizures, headache, confusion, and changes in vision

## **Class Effects:**

Class effects are potential risks that are associated with a particular group of drugs. Niraparib belongs to the group known as poly (ADP-ribose) polymerase inhibitors (PARP) inhibitors. These class effects are potential risks for the group of drugs but have not yet been identified as side effects for niraparib.

#### Secondary Primary Malignancy:

• PARP inhibitors may also cause a new primary cancer (that is, a cancer other than the one for which you have been treated). In 2 studies comparing niraparib to placebo (sugar pill), new primary cancers were observed in a small number of patients who took niraparib or placebo.

## **Side Effects Requiring Immediate Medical Attention:**

The side effects listed below require <u>IMMEDIATE MEDICAL ATTENTION OR ADVICE</u>. The study team will monitor you for these symptoms. Call the study doctor or the emergency contact on the first page of this form right away if you have any of these side effects:

- Symptoms of severe allergic reaction: Difficulty breathing, shortness of breath, low blood pressure (feeling lightheaded, dizziness), tingling around the mouth, or rash
- Symptoms of low platelet count: Bleeding and bruising
- Symptoms of low red blood cell count: tired or short of breath
- Symptoms of severe and life-threatening infection resulting from low neutrophil counts: Fever, feeling of low blood pressure (lightheadedness, dizziness), decreased urination, rapid pulse, rapid breathing or shortness of breath
- Decrease in the number of all types of all blood cells (pancytopenia)

Version: 1/21/2025 10 of 27

- Symptoms of a severe increase in blood pressure: Blurry vision, headache, nausea, vomiting, confusion, passing out, seizures, weakness or numbness on one side of body or in one arm or leg and/or difficulty talking (symptoms of a stroke), trouble breathing, chest pain, pain in the upper or lower back, urine that is brown or bloody
- Symptoms of neurological side effect from niraparib treatment: headache, vision changes, confusion or seizure with or without high blood pressure

## Safe Handling:

Niraparib may have adverse effects on an unborn baby. Wash your hands after handling the Study Drug. If a caregiver is giving the Study Drug to you, he or she should wear disposable gloves. Notify your Study Doctor if it appears that the Study Drug is damaged or defective in any way.

## <u>Ipilimumab</u>

Some of the side effects of ipilimumab may not cause you any symptoms, including changes in your liver or kidney function, changes in your thyroid, pituitary or adrenal gland function, changes in your blood count or changes in your electrolytes (salt levels in the blood). These will be assessed by the physician with blood tests at every treatment visit.

## **COMMON, SOME MAY BE SERIOUS**

In 100 people receiving ipilimumab more than 20 and up to 100 may have:

- Diarrhea
- Swelling and irritation of the colon (colitis)
- Increase in liver enzymes
- Fatique
- Skin itchiness
- Skin rash
- Nausea
- Abdominal pain
- Decreased appetite
- Fever
- Vomiting
- Headache
- Constipation
- Adrenal gland abnormalities, which may make you feel tired or make your blood pressure go down
- Thyroid gland abnormalities, which may make you feel tired or cold

## OCCASIONAL, SOME MAY BE SERIOUS

In 100 people receiving ipilimumab from 4 to 20 may have:

- Chills
- Weakness
- Muscle pain

Version: 1/21/2025 11 of 27

· Redness of skin

## RARE, AND SERIOUS

In 100 people receiving ipilimumab 3 or fewer may have:

- Decrease or total loss in hormones of the pituitary gland, which may make you feel tired
- Allergic reactions
- Irritation of the liver
- Irritation and swelling of the pituitary gland, which may give you a headache
- Decreased red blood cells, which may make you feel tired or dizzy
- · Loss of color (pigment) from areas of skin
- Decreased or blurry vision, or inflammation of the eye
- Numbness or tingling in your fingers or toes
- Inflammation or loss of the lining of the brain or spinal cord which may make you feel confused or give you a headache
- Inflammation of the kidneys
- Joint pain
- Pneumonitis

Death resulting from side effects considered related to ipilimumab occurred in about 1% of patients treated with ipilimumab in earlier clinical trials. Severe infections including sepsis have also been reported in ipilimumab-treated subjects, some of which resulted in death.

Our prior research does not suggest that combining ipilimumab plus niraparib increases the risk of either drug.

#### Other Study Related Risks

#### Risks of Using Up Stored Tumor Tissue Samples

If it is available, stored tumor tissue may be collected. It is possible that this entire stored sample will be used for the purposes of this research study and therefore may not be available for future clinical assessments as part of your routine care.

## Risks of Biopsy

A biopsy is an invasive test in which your cells and/or tissue are collected for examination. It involves the surgical removal of a small bit of tissue for examination. The biopsies may require image-guidance. Your study doctor will explain this procedure to you in more detail, and you will be given a standard hospital consent form to sign detailing your specific type of biopsy prior to the procedure.

#### Likely risks:

- Pain
- Discomfort
- Soreness
- Minor bleeding

Version: 1/21/2025 12 of 27

#### PARPVAX2

Bruising

#### Less likely risks:

- Redness
- Swelling
- Bleeding
- Pneumothorax (collapsed lung)

#### Rare risks:

- Bleeding, life threatening hemorrhage
- Possible damage to adjacent organs
- · Drainage from the biopsy site
- Abnormal wound healing
- Fever
- Infection
- Allergic reaction to the medication used to numb the skin over the biopsy site

#### **Blood Samples:**

There may be side effects of having blood drawn such as:

- Fainting
- Redness
- Pain
- Bruising
- Bleeding
- Infection
- Blood clots, which may cause inflammation, swelling and pain

If you feel faint tell the study staff right away.

## Risks of IV

An IV line will be used to administer study drug through a vein in your arm. The use of an IV line may cause discomfort, irritation, mild bruising, bleeding, leakage of drug solution, and rarely infection, nausea, and lightheadedness.

#### Risks of Infusion-Related Reaction

Infusions of drugs can cause allergic reactions in people. Allergic reactions may include shortness of breath, itching, rash, low blood pressure, and fever during the infusion or shortly after. If you experience any of these symptoms, you should contact your doctor immediately. Sometimes these reactions can be serious and can result in death if not watched carefully. You will be watched by medical personnel for signs of allergic reactions, and you will be given medicine if you need it.

#### Risks of Radiology Tests

During your participation in this study, you may undergo routine radiology tests to assess your disease.

Version: 1/21/2025 13 of 27

These can include CT, MRI, x-ray or PET/CT scans. Each of these procedures has risks associated with it, and you should talk to your study doctor or the person doing these procedures about the risks before they start.

- Radiation Exposure: This research study involves exposure to radiation from the CT scans, PET scans, x-rays, and image-guided biopsies. Therefore, you will receive a radiation dose. Some of these procedures may not be necessary for your medical care and will occur only as a result of your participation in the study. At doses much higher than you will receive, radiation is known to increase the risk of developing cancer after many years. At the doses you will receive, it is very likely that you will see no effects at all.
- CT Scans: A CT scan is an imaging method that uses x-rays to create cross-sectional pictures of the body. You will be asked to lie on a narrow table that slides into the center of the CT scanner. Depending on the study being done, you may need to lie on your stomach, back, or side. Once you are inside the scanner, the machine's x-ray beam rotates around you. It is important to remain still during the exam, because movement causes blurred images. You may be told to hold your breath for short periods of time. The scans take about 15 minutes or less to complete.
  - It is important to inform your study doctor if you have had an allergic reaction to IV contrast material in the past, or if you have an allergy to iodine. Most CT contrast reactions (approximately 95%) are mild to moderate in degree and most resolve themselves without treatment. However, life-threatening reactions and fatalities, mostly of cardiovascular origin, have occurred. People with heart disease, kidney disease or allergies are more likely to have a more severe reaction to contrast agents. If you have a history of kidney disease, allergies or heart disease, please inform the study staff. Likely contrast reactions include feelings of overall warmth (especially in the bladder area after injection), a metallic taste during the injection, and warmth, burning sensation, or momentary pain during the contrast injection at the injection site. Less likely contrast reactions include nausea, vomiting, headache, hives, and itching. Rare but serious contrast reactions include faster than normal heart rate (tachycardia), high blood pressure (hypertension), low blood pressure (hypotension), heart attack, kidney failure, fluid in the lungs (pulmonary edema), serious allergic reaction, and death. There is also a risk that multiple needle sticks will be necessary to ensure proper intravenous line placement. There may be a small amount of pain or bruising with the placement of the intravenous catheter (IV) and a small risk of infection at the injection site.
- MRI: The known risks associated with an MRI are minimal. The procedure uses radio waves and a magnetic field to take pictures. The greatest risk of having an MRI is the chance of metal objects flying through the air toward the magnet and hitting you. To reduce this risk, all people involved with the study are instructed to remove all metal from their clothing and all metal objects from their pocket. You must tell your study doctor if you have any metal plates or clips in your body. No metal objects are allowed to be brought into the magnet room at any time. Metal objects inside your body can affect the test results and could lead to injury. Because the magnetic field of the MRI scanner attracts metal, these studies will not be performed on anyone with a pacemaker or any non-removable metallic foreign objects in their body. If you have any such object on your body,

Version: 1/21/2025 14 of 27

you will not receive the scan. You may feel claustrophobic (fear of being closed in) or anxious. You may experience some discomfort and fatigue from lying in a confined space. There are no known effects from exposure to the magnetic fields. Multiple needle-sticks may be necessary if a vein cannot be properly accessed and this will be carried out upon your permission. It is possible that during the course of the research study, the research staff may notice an unexpected finding(s). Should this occur, the finding(s) will be considered by the appropriate personnel and the PI will inform you if necessary. These possible finding(s) may or may not be significant and may lead to anxiety about your condition and to further work-up by your physician.

PET/CT Scan: A PET scan is a type of imaging test that helps doctors see how the organs and
tissues inside the body are actually functioning. The test involves injecting a very small dose of a
radioactive chemical, or radiotracer, into a vein. Although a radiotracer chemical is used in this
test, the amount of radiation exposure is low. The dose of tracer used is so small that it does not
affect the normal processes of the body. The CT portion also gives a small radiation exposure. You
may experience discomfort related to lying still for a prolonged period of time.

## What about pregnancy and breastfeeding?

#### Reproductive Risks:

<u>Study drugs may have adverse effects on an unborn baby</u>. Study participants of reproductive potential must adhere to contraception (methods or ways to prevent pregnancy) requirements.

Effects of niraparib on fertility are unknown at this time. Animal studies in a drug similar to niraparib have been shown to cause a decrease in the number of cells that produce eggs in women's ovaries (reproductive organs).

Animal studies have shown that niraparib can cause a reversible decrease in sperm count. If you agree to participate in this study, you are expected to inform your female sexual partner(s) that you are participating in a clinical research study of an investigational drug, and that the effects of the drug on human sperm, an unborn baby and on a pregnant woman are unknown. You are also expected to provide your female sexual partner(s) with the information on the acceptable birth control methods described by your Study Doctor and to provide her with contact information for the Study Doctor for any additional questions. If your female partner becomes pregnant while you are participating in this study or within 90 days after your last dose of Study Drug, tell your Study Doctor right away as the Study Doctor is required to follow up and document the course and the outcome of all pregnancies. The Study Doctor may seek the pregnant woman's permission to review her medical records and the infant's medical records up to delivery, if applicable. The Study Doctor will share the information about your pregnant partner and the baby with the Sponsor to help understand the effects, if any, that the Study Drug may have on the pregnancy and/or the baby.

#### Female Participants

You should not become pregnant while on this study and for 6 months after your last dose of study drug because the study drugs could have a negative effect on an unborn baby. In addition, you should not breastfeed while on this study as these drugs may also affect a breast-feeding child. People who are Version: 1/21/2025

pregnant or breast-feeding (including expressing breastmilk for bottle feeding or storage) are not allowed to participate in this study. If you become pregnant, you will no longer be able to participate in this study.

If you are able to have children, you must agree to use two medically accepted forms of birth control including condoms, diaphragms, cervical cap, an intra-uterine device (IUD), intrauterine hormone-releasing system (IUS), surgical sterility (tubal ligation or a partner that has undergone a vasectomy), or oral, injectable, or implantable contraceptives, OR you must agree to completely abstain from intercourse during participation in this study and for 6 months after your last dose of study drugs. Abstinence at certain times of the cycle only, such as during the days of ovulation, after ovulation and withdrawal are not acceptable methods of birth control. Your study doctor must approve your form of birth control. Ask your study doctor about the contraceptive methods that are available and which might be the best for you.

Even when you use an approved contraceptive method, there is always a small risk that you could still become pregnant. If you do become pregnant during the course of this study, or up to 6 months after your last dose of study drug, you must discontinue study treatment, tell the investigator immediately, and consult an obstetrician or maternal-fetal specialist. If you become pregnant while on this study, we will ask permission to collect information about your pregnancy.

• Tell the study doctor if you are pregnant. If you get pregnant during the study, you will not receive any more niraparib, but you may remain in the study for follow-up. You must not breastfeed an infant (or store breastmilk for use) while taking the Study Drug and for 30 days after receiving final dose of Study Drug. We will follow-up until the delivery of the baby.

#### Male Participants

To participate in the study, male study participants must adhere to contraception (methods or ways to prevent pregnancy) requirements.

You should not father a child or donate sperm while on this study and for 90 days after your last dose of study drug, because the drug involved could have a negative effect on an unborn baby. If your spouse or partner has the potential to become pregnant, you and your partner must use two medically accepted forms of birth control including condoms, diaphragms, cervical cap, an intra-uterine device (IUD), intrauterine hormone-releasing system (IUS), surgical sterility (tubal ligation or a partner that has undergone a vasectomy), or oral, injectable, or implantable contraceptives, OR you must agree to completely abstain from intercourse during participation in this study and for 90 days after your last dose of study drugs. Abstinence at certain times of the cycle only, such as during the days of ovulation, after ovulation and withdrawal are not acceptable methods of birth control. Your study doctor must approve your form of birth control. Ask your study doctor about the contraceptive methods that are available and which might be the best for you.

You should also inform your partner of the potential harm to an unborn child. She should know that if a pregnancy should occur during the course of this study, or up to 90 days after your last dose of study drug, you will need to report it to the study doctor immediately, and she should promptly notify her doctor. The study doctor will also ask to follow-up on the pregnancy.

Version: 1/21/2025 16 of 27

#### Genetic Research Risks:

As part of this research study, the study team may perform genetic testing on your tumor and/or blood samples. These are experimental tests, not approved by the FDA, and will have no impact on your study participation. Results will not appear in your medical record and your doctor will not be notified directly. New health information about inherited traits that might affect you or your blood relatives could be found during the research study. Even though your genes are unique, you share some of the same genes with your blood relatives. Although we are not able to know all of the risks from taking part in research on inherited traits, we believe the risks to you and your family are very low, because your samples will be coded.

Very rarely health or genetic information could be misused by employers, insurance companies, and others. For example, life insurance companies may charge a higher rate based on this information. The chance that your information could be misused is very small. We have many protections in place to lower this risk. Your privacy will be protected to the fullest extent possible.

A new federal law called the Genetic Information Non-Discrimination Act, or GINA is in effect. This law helps to lower the risk of health insurance or employment discrimination. The law does not include other types of misuse by life insurance or long term care insurance. To learn more about the GINA Law, please check the Internet or ask the study staff.

## What happens if we find a gene that might predispose you to getting cancer?

The genetic testing done as a part of this study is purely experimental. The results of these tests will not be included in your medical record. If during this experimental testing we identify a mutation in a gene that we think might predispose you to getting cancer, we will notify you of this finding. If you would be interested at that time in having clinical genetic counseling and confirmatory testing done, we can offer those services to you. Only the results of any clinical genetic testing you might choose to have done would be made a part of your medical record. A separate consent form that you will be given specifically for clinical genetic testing will explain in detail that testing and how the results may be used.

In the event we identify a gene mutation and you cannot be contacted, you may indicate the name and contact information of the person we may release this information to at the end of this form.

# What if new information becomes available about the study?

During the course of this study, we may find more information that could be important to you (such as new information about how the drug works or newly discovered side effects). If we discover new information about the study that could affect your decision to stay in the study, you will be notified in a timely manner. You will be able to ask questions about this new information and can discuss it with your family, friends, or doctor.

# What are the possible benefits of the study?

Taking part in this study may or may not make your health better. However, while you may not benefit

Version: 1/21/2025 17 of 27

personally, the knowledge learned from your participation in this research study may benefit other patients in the future. It is possible that your disease and/or health may worsen as a result of participating in this study.

## What other choices do I have if I do not participate?

Your participation in this study is entirely voluntary. Other possible options include:

- Getting treatment or care for your cancer without being in a study. This would include chemotherapy such as FOLFIRI
- Taking part in another study.
- Not receiving treatment at this time.
- Getting comfort care, also called palliative care. This type of care helps reduce pain, tiredness, appetite problems and other problems caused by the cancer. It does not treat the cancer directly, but instead tries to improve how you feel. Comfort care tries to keep you as active and comfortable as possible.

Talk to your doctor about your choices before you decide if you will take part in this study.

## Will I be paid for being in this study?

You will not be paid for taking part in this study and you will not receive reimbursement for travel expenses.

## Will I have to pay for anything?

The drug manufactures, GSK and BMS, will supply the study drugs, Niraparib and Ipilimumab, at no charge while you take part in this study. The cost of drug administration may be the responsibility of you and/or your insurance provider.

You will be responsible for any deductibles or applicable co-pays for the standard tests, exams or procedures that would be done for your routine clinical care, such as office visits, scans and blood work. You and/or your insurance provider will be responsible for standard tests, exams or procedures that would be done even if you were not in this study. Please talk to your doctor and study team about putting you in touch with a financial counselor to determine exactly what the deductible and co-pay will be for you; this is highly variable depending on your type of insurance. There will be no charge to you for those laboratory tests and other procedures that are being done specifically for the purposes of this research study.

For more information on clinical trials and insurance coverage, you can visit the National Cancer Institute's Website at: http://cancer.gov/clinicaltrials/understanding/insurance-coverage. You can print a copy of the "Clinical Trials and Insurance Coverage" information from this Website.

Another way to get the information is to call 1-800-4-CANCER (1-800-422-6237) and ask them to send you a free copy.

# What happens if I am injured or hurt during the study?

If you have a medical emergency during your participation on this study, you should go to the nearest emergency room. If you think you have been injured as a result of taking part in this Study, you should

Version: 1/21/2025 18 of 27

contact the Principal Investigator or Emergency contact listed on page one of this form as soon as possible. You may also contact your own doctor, or seek treatment outside of Penn Medicine. Be sure to tell the doctor or his/her staff that you are in a research study being conducted at Penn Medicine. Ask them to call the telephone numbers on the first page of this consent form for further instructions or information about your care.

Penn Medicine will also offer you the care needed to treat side effects and/or injuries that occur while you are taking part in this research.

We may bill your insurance company or other third parties, if appropriate, for the costs of the care you get for any injury. You may also be responsible for some of these costs. There are no plans for Penn Medicine, Lusgarten Foundation, BMS or GSK to pay you or give you other compensation for the injury. You do not give up your legal rights by signing this form.

You may receive bills for side effects/injuries that occur during your participation in this study. If you have questions about these bills and whether or not they are covered by the research study, please bring copies of these bills to a member of the study team and they will be able to answer your questions.

## When is the Study over? Can I leave the Study before it ends?

This study is expected to end after all participants have completed all visits, and all information has been collected. This study may also be stopped at any time by the Principal Investigator, sponsor or the Food and Drug Administration (FDA) without your consent because:

- The Primary Investigator feels it is necessary for your health or safety. Such an action would not require your consent, but you will be informed if such a decision is made and the reason for this decision.
- You have not followed study instructions, or you become pregnant
- The Sponsor, the study Principal Investigator, or the Food and Drug Administration (FDA) has decided to stop the study due to new information regarding side effects.
- For any other reason that is not known at this time.

If you are removed from the research study, your study doctor will explain to you why you were removed. The study doctor and study team will help arrange for your continued care.

If you decide to participate, you are free to leave the study at any time. Withdrawal will not interfere with your future care.

# How will my personal information be protected during the study?

If you decide to participate in this study, the study doctor and staff will collect medical and personal information about you as part of completing the study. We will do our best to make sure that the personal information in your medical record will be kept private. However, we cannot guarantee total privacy. Your personal information may be given out if required by law. If information from this study is published or presented at scientific meetings, your name and other personal information will not be used. This study is being overseen by the Food and Drug Administration (FDA); therefore, they may review your research records. Please refer to the information below which explains more specifically how your personal information will be protected. If you do not want to allow these uses, you should not participate in this Version: 1/21/2025

study. Information identifying you will be kept confidential as described below.

While collected as part of this study by your study doctor and study team, identifying information (including, but not limited to, your name, address, telephone number, medical record number, or any number/codes that will directly identify you) will be kept as confidential as possible and will not be routinely disclosed outside of Penn Medicine. Personal health information that could be used to identify you will not routinely be sent to Lustgarten Foundation, the drug manufactures, BMS and GSK, and/or their designated representatives.

You will be assigned a unique subject registration number upon enrollment. This number and your initials will be used to identify you throughout the course of this study so that your identity is protected. The key to this code (which links your name back to the personal health information collected during this study) will be stored in a secure area and only the Penn Medicine study team will have access to this code. However, some of the study data (e.g. date of birth) could be used in combination with other information, in order to identify you. If you have questions about the specific information that will be released, you should ask your study doctor.

If you test positive for HIV, by law we have to report the positive test results to the City of Philadelphia Health Department and/or the PA Department of Health. Personal identifiers such as name, sex, date of birth, address, and phone number will be reported. For more information about the requirements reporting infectious diseases to the City of Philadelphia Health Department, please visit <a href="https://hip.phila.gov/ReportDisease">https://hip.phila.gov/ReportDisease</a>. For more information about the requirements reporting infectious diseases to the PA Health Department, please visit <a href="https://www.health.pa.gov">https://www.health.pa.gov</a> and type 'Reportable Diseases' into the site search bar.

# Will information about this study be available to the public?

A description of this clinical trial will be available on <a href="http://www.ClinicalTrials.gov">http://www.ClinicalTrials.gov</a>, as required by U.S. Law. This Web site will not include information that can identify you. At most, the Web site will include a summary of the results. You can search this Web site at any time.

# What may happen to my information and samples collected on this study?

#### Collection of Identifiable Specimens

Your samples may be used to create products, including some that may be sold and/or make money for others. If this happens, there are no plans to tell you, or to pay you, or to give any compensation to you or your family.

Whole genome sequencing may be conducted on your samples. Whole genome sequencing involves analyzing your entire personal genetic code. WGS can be conducted to determine changes and mutations in DNA. The significance of these results may not be well defined. Not all genetic variations affect one's health.

#### Future Use of Data and/or Specimens

Your identifiable information will be stored indefinitely and may be used for future research purposes. If you consent to the optional storage of your samples for future research, your samples will be stored

Version: 1/21/2025 20 of 27

indefinitely or until used up. If you do not consent to the optional storage of your samples for future research, your sample will be destroyed at the end of the study. Future researchers may receive information that could identify you. This can be done without again seeking your consent in the future, as permitted by law. The future use of your information and samples only applies to the information and samples collected on this study.

The following identifiers will be retained with your information and samples: the information and samples will be labeled with your study ID. The study ID is linked back to your identifiable information (i.e. the master list).

Your information and samples may be stored and used for future research purposes for an indefinite amount of time. Samples will be stored for future use only if you agree at the bottom of the form.

There are no plans to tell you about any of the specific research that will be done. Possible future research may include additional studies that further characterize tumor and host factors that may influence response and resistance to treatment.

We may share your identifiable information and samples with other researchers within Penn, or other research institutions as well as pharmaceutical, device, or biotechnology companies that may develop genomic (DNA- or RNA-based) signatures. We will not follow up with you to tell you about the specific research that will be done. We will not give you any results from these studies. It is possible that you may have chosen not to participate in these future research studies, had you been approached for participation. You will not be given the results from testing that may be performed on your identifiable specimens as part of future research.

There is a risk of breach of confidentiality (unintentional release of your information). We will do our best to make sure that this doesn't happen. However, we cannot guarantee total privacy. We will protect your confidentiality during storage and sharing by not releasing identifiable information. Your information and samples will be labeled with a code that links you to the information (i.e. master list), but we will not share the master list.

You will likely not directly benefit from future research with your information and samples. Research with your identifiable information and samples may help others by improving our understanding of health and disease, improving health care and making safer or more effective medical therapies, and developing new scientific knowledge.

If you have questions about the storage of your information and samples, or have changed your mind, you can contact Dr. Reiss at 215-360-0735. If you change your mind, you can ask to have the data collected about you removed or the samples destroyed. You can also ask us to remove information that identifies you from the data or samples. However, this may not be possible if your samples and data have already been shared.

# **Electronic Medical Record and Release of Study Related Information?**

#### What is an Electronic Medical Record?

An Electronic Medical Record (EMR) is an electronic version of your medical chart within a health system. An EMR is simply a computerized version of a paper medical record.

Version: 1/21/2025 21 of 27

If you have never received care within Penn Medicine and are participating in a Penn Medicine research study that uses Penn Medicine healthcare related services, an EMR will be created for you for the purpose of maintaining any information produced from your participation in this research study. The creation of this EMR is required for your participation in this study. In order to create your EMR, the study team will need to obtain basic information about you that would be similar to the information you would provide the first time you visit a hospital or medical facility (i.e. your name, the name of your primary doctor, the type of insurance you have). If you have been a patient at Penn Medicine in the past, information from your research participation will be added to your existing medical record.

## What may be placed in the EMR?

Information related to your participation in the research (e.g., laboratory tests, notes from your physician, imaging studies, and clinical procedures, etc.) will be placed in your EMR maintained by Penn Medicine.

Once placed in your EMR, your information may be accessible to appropriate Penn Medicine workforce members that are not part of the research team. Information within your EMR may also be shared with others who are determined by Penn Medicine to be appropriate to have access to your EMR (e.g. health insurance company, disability provider, etc.).

Penn Medicine also participates in automated information sharing through Health Information Exchanges (HIEs). HIEs securely share parts of your electronic health record, including research information, with other healthcare organizations involved in your care. This information is shared to improve the quality, safety and efficiency of your healthcare. To request that your health information not be shared through HIEs, please call 215-662-4484.

#### Will I, as a subject, have access to research related information within the EMR?

The 21<sup>st</sup> Century Cures Act requires healthcare institutions to allow patients increased access to their electronic medical record. As part of your participation in this research, you will have access to research related information within your EMR through Penn Medicine's patient portal- called MyPennMedicine (MPM).

Some research results may be placed in your medical record. For example, the results from testing conducted in a laboratory or center that is part of Penn Medicine for standard medical tests/procedures aligned with routine care (vital signs, blood work such as chemistry/hematology testing, and tumor imaging) will be entered in your medical record. This would be done regardless of research participation. Results placed in the medical record are part of the designated record set and you have a right to review these results per HIPAA regulations. For these types of research results, you will be notified of your returned results in a timely manner, without delay, in the same way you would if not participating in this research.

Other research results will not be placed in your medical record. For example, the results from the biospecimen testing conducted in a laboratory that is not part of Penn Medicine and/or results from testing conducted in a noncertified laboratory (i.e., the results would not have been placed in the medical record as part of clinical care) will not be entered in your medical record. You will not have access to these results through your medical record as these results are returned only in the research database.

Version: 1/21/2025 22 of 27

## Will I receive the results of research testing that may be relevant to my health?

Clinically relevant research results will be disclosed to you; this will be done in the context of discussion with your study doctor and/or clinical treatment team. Results from clinical testing done as part of this research will be placed in your medical record. Results placed in the medical record and will be available to you per HIPAA regulations, as noted above.

## What information about me may be collected, used or shared with others?

The following personal health information will be collected and used for the purposes of this study.

- Name, address, telephone number, email address, date of birth
- The history and diagnosis of your disease
- Specific information about the therapy you received, including previous treatment(s) you may have had
- Information about other medical conditions that may affect your care
- Medical data including laboratory test results, health status, EKGs, CTs, x-rays, MRIs, PETs, pathology results, etc.

- Information on side effects (adverse events) you may experience, and how these were treated
- Long-term information about your general health status and the status of your disease. This may include information from other health care providers.
- Data that may be related to tissue samples that may be collected from you
- Numbers or codes that will identify you, such as your medical record number and/or Medicare ID number
- Information related to study visits and other tests/procedures performed while you are participating on this study.

# Why is my personal health information being used?

Your personal contact information is important for the research team to contact you during the study. For this study we may need to contact you via email to provide you information about scheduling, appointments, notes or to send you information about your participation in the study. Email communications are often not secure and may be seen by others as a result. By signing below, you accept this risk. If you wish for us to use a different means to communicate with you during the course of this study please discuss this with the research team and alternative methods can be arranged.

Your personal health information and results of tests and procedures are being collected as part of this research study, and will be used to conduct and oversee this research study, and to help guide your medical care.

# Where may my information be stored?

Information related to your participation in clinical research will be contained in a clinical research management system (CRMS) at Penn Medicine. A clinical research management system (CRMS) is used to register your information as a participant in a study. This allows for your research data to be entered and stored for the purposes of study operational and financial applications and other activities required as part Version: 1/21/2025

of the conduct of the research. Once placed in the CRMS your information may be accessible to other authorized personnel at Penn Medicine that support research operations.

Your de-identified information will be held in the Lustgarten United Clinical Information Database (LUCID). LUCID is a data depository created by the sponsor of this study, the Lustgarten Foundation. In LUCID, you will not be identified by name, medical record number, address, telephone number, or any other direct personal identifier.

Your information may be held in other research databases.

## Who can see or use my information?

Which Penn Medicine personnel may use or disclose my personal health information?

The following individuals may use or disclose your personal health information for this research study:

- The Principal Investigator and the Investigator's study team
- Authorized members of the workforce of Penn Medicine, and Penn Medicine support offices, who
  may need to access your information in the performance of their duties (for example: for research
  oversight and monitoring, to provide care as part of this study or as part of your routine care, to
  manage accounting or billing matters, etc.). This includes members of the Institutional Review
  Board (IRB), an Ethics Committee at Penn Medicine who are responsible for reviewing and
  overseeing research studies to ensure that they are safe and being well managed.
- Other research personnel with access to the databases for research and/or study coordination and as otherwise approved by the IRB

#### Who, outside of Penn Medicine, might receive my personal health information?

As part of the study, the Principal Investigator, the study team and others listed above, may disclose your study-related records, including the results of the research study tests and procedures, to those listed below. This study data may be processed and transmitted using secure computer systems. In all disclosures outside of Penn Medicine, you will not be identified by name, medical record number, address, telephone number, or any other direct personal identifier unless disclosure of the direct identifier is required by law. In records and information disclosed outside of the Penn Medicine, you will be assigned a unique code number.

Your original medical records also may be reviewed by the sponsor of this study or its designated representatives, the Institutional Review Board overseeing this study, and any of the regulatory or safety oversight organizations outlined below. They may review these records for the purpose of checking data collected for the study, to make sure the study is being done properly, and to analyze the results of the study.

Research data generated from your participation in this study will be de-identified and deposited in the sponsor's database, LUCID. The de-identified data in LUCID will be made available to the sponsor of this study and its designated representatives for purposes of research.

Version: 1/21/2025 24 of 27

## Individuals or organizations responsible for administering the study:

- Lustgarten Foundation (the sponsor of this study) and their designated representatives
- BMS and their designated representatives
- GSK and their designated representatives
- · Penn Medicine and Kim A. Reiss, MD
- Dana Farber Cancer Institute and Brandon Huffman, MD

#### Regulatory and safety oversight organizations

- The U.S. Food and Drug Administration (FDA)
- Office for Human Research Protections (OHRP)
- Other regulatory agencies and/or their designated representatives, including international agencies
- Public Health agencies and other government agencies (including non-U.S.) as authorized or required by law

Once your personal health information is disclosed to others outside of Penn Medicine, it may no longer be covered by United States federal privacy protection regulations.

The Principal Investigator or study staff will inform you if there are any additions to the list above during your active participation in the trial. Any additions will be subject to Penn Medicine procedures developed to protect your privacy.

#### How long may Penn Medicine be able to use or disclose my personal health information?

Your authorization for use of your personal health information for this specific study does not expire. If you sign this form, we will collect your health information until the end of the research study. We may collect some information from your medical records even after you finish taking part in this study or after your death. We will keep all of the information forever in case we need to look at it again. We will protect this information and keep it confidential.

Your information may be held in a research database. However, Penn Medicine may not re-use or redisclose information collected in this study for a purpose other than this study unless:

- You have given written authorization to do so
- Penn Medicine's Institutional Review Board grants permission after ensuring that appropriate privacy safeguards are in place
- As permitted by law

The data from this study may be published or used for teaching purposes, however you will not be personally identified in any publication. Your identity will remain confidential unless disclosure is required by law.

#### What if I decide not to give permission to use and give out my health information?

Then you will not be able to be in this research study.

Version: 1/21/2025 25 of 27

## Can I change my mind?

You have the right to withdraw your permission for the use of your personal health information, but if you do so, you must stop taking part in this study. You must do so in writing to the Principal Investigator at the address on the first page. Even if you withdraw your permission, your personal health information that was collected before we received your written request may still be used and disclosed, as necessary for the study. If you withdraw your permission to use your personal health information, you will also be withdrawn from the research study and no new information will be collected. However, even if you do withdraw your permission to use the data about you, we are required by the FDA and other national regulatory authorities to record anything that relates to the safety of the investigational drug under study.

#### Will I be able to access my research records?

You have the right to see and get a copy of your medical records kept by Penn Medicine. However, you will not be able to review or receive some of your records related to the study until after the entire study has been completed. When the study is over, you may write to the study doctor to ask to see or copy all of your medical information that was collected during the study. You also have the right to say how your medical information may be used, and to have any incorrect data about yourself updated or corrected.

By signing this document, you are permitting the Penn Medicine to use and disclose personal health information collected about you for research purposes as described above.

# Who can I call with questions, complaints or if I'm concerned about my rights as a research subject?

If you have questions, concerns or complaints regarding your participation in this research study you should speak with the Principal Investigator listed on page one of this form. If you have any questions about your rights as a research subject, you may contact the Office of Regulatory Affairs at the University of Pennsylvania with any questions, concerns or complaints by calling (215) 898-2614.

# Where can I get more information?

You may call the National Cancer Institute's Cancer Information Service at 1-800-4-CANCER (1-800-422-6237). You may also visit the NCI website at http://cancer.gov/. For NCI's clinical trials information, go to http://cancer.gov/clinicaltrials/. For NCI's general information about cancer, go to http://cancer.gov/cancerinfo.

Version: 1/21/2025 26 of 27

# **Making Your Decision**

Please circle "yes" or "no" below and initial next to your choice to indicate whether or not you agree to participate in the optional research:

| 1. I consent to the storage of my blood for use now and for future research: | | | | |
|---|---|---|---|---|
| Yes No Initials: 2. I consent to the storage of my tumor tissue for use now and for future research: | | | | |
| Yes | No | Initials: | | |
| When you sign this form, you are agreeing to take part in this research study. This means that you have read the consent form, the study has been explained to you, your questions have been answered, you have had time to make your decision, and you have decided to volunteer to participate. You have been given the names of study staff that you can contact if you need assistance or if you have any additional questions or concerns. You agree to follow all of the instructions of your study doctor to the best of your ability, and report any changes in your health that may occur during the study. | | | | |
| Your signature also means that you are permitting Penn Medicine to use your personal health information collected about you for research purposes within our institution. You are also allowing Penn Medicine to disclose that personal health information to outside organizations or people involved with the operations of this study. | | | | |
| You agree | that your primary care | e physician can be info | ormed about you | ur participation in this clinical trial. |
| A copy of the | nis signed and dated co | onsent form will be giv | en to you. | |
| Name of F | Participant (Print) | Signature of Partic | pant | Date |
| Name of F<br>Authorizat | Person Obtaining ion (Print) | Signature of Perso<br>Authorization | n Obtaining | Date |

Version: 1/21/2025 27 of 27